CLINICAL TRIAL: NCT01661738
Title: Phase II Clinical Trial of Group ACYW135 Meningococcal Polysaccharide Vaccine
Brief Title: Clinical Trial of Group ACYW135 Meningococcal Polysaccharide Vaccine 002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hualan Biological Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hualanbio-Meningococcal CT 002; Hualanbio-phase II CT (Other Grant/Funding Number: Hualan Biological Engineering Inc.)
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Meningitis
Keywords: Group ACYW135 Meninigococcal Polysaccharide Vaccine
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group ACYW135 Meningococcal Polysaccharide Vaccine (Experimental): 0.5 ml/ vial
  Interventions: Biological: Group ACYW135 Meningococcal Polysaccharide Vaccine

INTERVENTIONS:
Biological: Group ACYW135 Meningococcal Polysaccharide Vaccine — 360 subjects were divided into three groups (120 subjects in each group), children (2~6 years of age), early youth (7~15 years of age) and adult (16~30 years of age) to receive Group ACYW135 Meningococcal Polysaccharide Vaccine, 0.5 ml, one dose regime
  Other Names: Hualan Bio

SUMMARY:
The clinical trial was designed to evaluate the safety and immunogenicity against Group ACYW135 Meningococcal Polysaccharide Vaccine of Hualan administered on subjects 2 years of age and older.

DETAILED DESCRIPTION:
Complying with requirements of the approval letter of clinical trial issued by SFDA (Approval Letter No.: 2006L01017), Hualan conducted phase II clinical trial of Group ACYW135 Meningococcal Polysaccharide Vaccine to evaluate the safety and immunogenicity of the experimental vaccine.

The safety end points were the presence of any systemic, local and adverse reaction. Evaluation indicators of immunogenicity were bacteriocin levels of groups A, C, Y and W135 respectively in the serum after the whole vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy permanent residence 2 years of age and older, the subjects (or their guardians) are able to understand and sign the informed consent;
* Healthy male or female by oral history, physical examination and clinical judgment and who complies with vaccination of this product;
* Be able to comply with the requirements of clinical trial protocol and immunogenicity examination;
* Have no history of vaccination within the past 3 months and vaccination with other products within the last 2 weeks;
* Axillary temperature ≤37.0℃.

Exclusion Criteria:

* Any acute disease, such as: tumor, autoimmunity disease, progressive atherosclerotic disease or diabetes with complication, chronic obstructive pulmonary disease need oxygen uptake, acute or progressive hepatopathy or nephropathy, congestive heart-failure, etc.;
* Allergic to vaccines or drugs (history of allergy to any vaccine in the past);
* History of neurologic symptom or signs;
* Known or suspected (or high risk) impaired or abnormal immune function, e.g.: receive immunosuppressant or immunopotentiator therapy, take immunoglobulin or blood product or plasma extract (except the gastrointestinal tract) within the past 3 months, HIV infection or related disease, etc.;
* History of meningitis infection or vaccination of meningococcal vaccine within the past 3 months;
* History of receiving other vaccines or immunoglobulin injection or any research drugs;
* Any acute disease needing application of antibiotics or anti-virus treatment in the whole body within the past 1 week;
* History of fever within the past 3 days (axillary temperature ≥38.0℃);
* Participating in another clinical trial;
* History of allergy, eclampsia, epilepsy, encephalopathy and mental disease or family disease;
* Thrombopenia or other coagulopathy that may cause contraindication to intramuscular injection;
* Acute chronic disease (such as Down syndrome, diabetes, sickle cell anemia or neurologic disease, Guillain-Barre Syndrome);
* Known or suspected diseases, including: respiratory system disease, acute infection or active stage of chronic disease, SBAV infection of children or mothers, cardiovascular disease, acute hypertension, cancer treatment, skin disease, etc.;
* Pregnancy
* Any condition that, in the judgment of investigator, may affect trial assessment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety | Day 28 after vaccination
  Systemic and local adverse reactions after the vaccination; adverse events

SECONDARY OUTCOMES:
Immunogenicity | The 4th week after immunization
  4-fold (seroconversion) and 8-fold increase of bactericidin; GMT and bactericidin increase after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Fubao Ma, Bachelor, Principal Investigator — Immunization Program Institute of Jiangsu Provincial Center for Disease Control and Prevention